CLINICAL TRIAL: NCT03263364
Title: Genomic Screening for Hereditary Erythrocytosis and Related Diseases
Acronym: GENRED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: GIRODON PRTS 2015
Record Dates: First submitted 2017-08-23; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Hereditary Erythrocytosis/Idiopathic Erythrocytosis
MeSH Terms: conditions — Polycythemia, primary familial and congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Unexplained polycythemias are rare diseases, and therefore, the collection of data inherent to these diseases will not only improve their characterisation, but also allow stratification according to the risks and the course of the disease. The objective of this project is to constitute a database on the disease which will allow us to better understand it and in due course improve its management.

The GENRED project thus bears uniquely on the collection of information, which will be gathered throughout the usual management of patients for this type of disease.

ELIGIBILITY:
Inclusion Criteria:

The characteristics of the patients included in the database will be described in terms of numbers and percentages for qualitative variables and in terms of means and standard deviations or medians and interquartile intervals for quantitative variables.

Exclusion Criteria:

The first step will be to exclude acquired secondary (pulmonary, renal and cardiac) or acquired primary (polycythemia vera due to JAK2 mutations) causes. The family history and the determination of serum EPO levels are very useful in the decision regarding which molecular tests should be performed first.

* patients without absolute erythrocytosis (i.e. without an increased red cell mass >125% of mean predicted value, or if the haematocrit is <60% in males or <56% in females.
* erythrocytosis related to polycythemia vera according to the 2008 WHO (World Health Organization) criteria
* Secondary erythrocytosis related to an obvious cause (renal lesions, chronic lung or heart diseases, endocrine lesions, miscellaneous tumours producing EPO, drugs such as androgens, hepatic lesions…)
* Low venous blood p50: the determination of p50 (percentage at which Hb is half saturated with oxygen) is very helpful is establishing the presence of a haemoglobin variant with high oxygen affinity or a rare 2,3-diphosphoglycerate (2,3-DPG) deficiency. In such a situation, a specific HBB, HBA1 and HBA2 mutation will be screened for using Sanger sequencing (these genes are not included in NGS analysis because of redundancy of pseudogenes).

In order to rule out non-informative erythrocytosis cases, a form including mandatory further tests must be filled in for a selection step. The required tests are: complete blood counts

* Blood electrolytes
* Arterial and venous gazes
* Serum erythropoietin dosage
* Liver function tests
* JAK2 mutations (both V617F and exon 12)
* Bone marrow aspirate and/or biopsy and/or endogenous BFU-E culture
* Abdominal ultrasound
* Lung function tests

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hereditary Erythrocytosis/Idiopathic Erythrocytosis
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Germline mutations that cause Hereditary Erythrocytosis/Idiopathic Erythrocytosis | at baseline

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Dijon Bourgogne, Dijon
  - CHU de NANTES, Nantes